CLINICAL TRIAL: NCT00077077
Title: A Phase I Study Of The Combination Of Oral DJ-927 And Capecitabine In Patients With Advanced Solid Tumors
Brief Title: DJ-927 and Capecitabine in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000346368; DAIICHI-927A-PRT006; WSU-085503MP4F
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — tesetaxel; Capecitabine

INTERVENTIONS:
Drug: DJ-927
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as DJ-927 and capecitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of DJ-927 and capecitabine in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of DJ-927 and capecitabine in patients with locally advanced or metastatic solid tumors.
* Determine the dose-limiting and non-dose-limiting toxic effects of this regimen in these patients.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the possible pharmacokinetic interactions of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation, nonrandomized, multicenter study.

* Course 1: Patients receive oral DJ-927 once on day 1 and oral capecitabine once on days 0 and 1 and twice daily on days 2-14.
* Course 2: Patients receive DJ-927 as in course 1 and oral capecitabine twice daily on days 2-15.
* Course 3 and all subsequent courses: Patients receive DJ-927 as in course 1 and oral capecitabine twice daily on days 1-14.

All courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of DJ-927 and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients receive treatment at the MTD.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30-40 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor

  * Locally advanced or metastatic disease
* Minimally pretreated
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin no greater than 1.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Gastrointestinal

* No prior chronic diarrhea
* No swallowing and/or malabsorption problems
* No diarrhea (excess of 2-3 stools/day above normal frequency in the past month)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No prior severe or life-threatening hypersensitivity reaction to a taxane or capecitabine
* No concurrent serious infection
* No neuropathy grade 2 or greater
* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other severe or uncontrolled underlying medical disease that would preclude study participation
* No psychiatric disorder that would preclude giving informed consent or study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic therapy

Chemotherapy

* Recovered from prior chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Recovered from prior radiotherapy
* No concurrent anticancer radiotherapy

  * Concurrent localized radiotherapy to a non-indicator lesion for pain relief is allowed provided other methods of pain control are ineffective

Surgery

* At least 4 weeks since prior major surgery and recovered
* No prior major surgery in the stomach or small intestine

Other

* At least 4 weeks since prior myelosuppressive therapy
* More than 28 days since prior investigational drugs (including analgesics and/or antiemetics)
* No other concurrent anticancer therapy
* No other concurrent anticancer cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Takimoto, MD, PhD, FACP — Cancer Therapy and Research Center, Texas
Locations (3):
- United States (3):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Cancer Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Result] Saif MW, Sarantopoulos J, Patnaik A, Tolcher AW, Takimoto C, Beeram M. Tesetaxel, a new oral taxane, in combination with capecitabine: a phase I, dose-escalation study in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2011 Dec;68(6):1565-73. doi: 10.1007/s00280-011-1639-3. Epub 2011 May 6. PMID 21547572